CLINICAL TRIAL: NCT05123963
Title: Restoring 24-hour Substrate Rhythmicity to Improve Glycemic Control by Timing of Lifestyle Factors
Acronym: TIMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: University of Calgary (Other); University of Waterloo (Other); Laval University (Other); Wageningen University (Other); Maastricht University Medical Center (Other); Leiden University Medical Center (Other); McMaster University (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MP-31-2021-4011
Record Dates: First submitted 2021-10-14; First posted 2021-11-17 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Prediabetic State
Keywords: Postprandial metabolism; High-intensity interval training
MeSH Terms: conditions — Prediabetic State | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Two randomized groups in parallel (Exercise training in the morning versus exercise training in the evening). In each group, the protocol will be carried out as a within-subject in which each subject will serve as his/her own control (before/after acute or prolonged exercise).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning exercise (Active Comparator): Participant to perform high-intensity interval training in the morning (~9 am)
  Interventions: Behavioral: High-intensity interval training
- Afternoon exercise (Experimental): Participant to perform high-intensity interval training in the morning (~4 pm)
  Interventions: Behavioral: High-intensity interval training

INTERVENTIONS:
Behavioral: High-intensity interval training — 3 times per week high-intensity interval training (HIIT) on a cycle ergometer for 12 weeks.

SUMMARY:
Exercise is well-known to improve skeletal muscle energy metabolism and is an established intervention to improve muscle insulin sensitivity and to counter the development of type 2 diabetes (T2D). However, given the 24h rhythmicity in substrate metabolism previously observed in healthy, lean men and the lack of such rhythmicity in men with insulin-resistance, the investigator hypothesize that appropriate timing of exercise training can maximize the metabolic health effects of exercise. Indeed, a preliminary study in humans revealed that afternoon high-intensity interval training (HIIT) exercise was more effective than morning exercise in improving 24h blood glucose levels in men with T2D. Another recent study in mice showed that the time of day is a critical factor in augmenting the beneficial effects of exercise on the skeletal muscle metabolome as well as on whole-body energy homeostasis. However, human studies that specifically target the impact of timing of exercise training on glucose homeostasis and metabolic health are scarce and the potential underlying mechanisms largely unknown.

The overarching goals of this project is to improve 24-hour rhythmicity of metabolism in men and women with prediabtes by appropriate timing of exercise and to assess its effect on metabolic health and immune response. Acute and prolonged exercise interventions timed in the morning vs late afternoon will be carried out in individuals with prediabetes to determine whether acute exercise in the afternoon and prolonged exercise training in the afternoon can improve peripheral insulin sensitivity, compared to exercise in the morning, and positively affect adipose tissue dietary fatty acid storage and partitioning of dietary fatty acids in skeletal muscles.

DETAILED DESCRIPTION:
Three metabolic studies A, B and C using PET imaging will be carried out at the CRCHUS. The 12-week exercise training intervention will consist of supervised cycling high-intensity interval training (i.e. short bouts of high-intensity exercise interspersed with short periods of rest) every other day at the CRCHUS. Continuous glucose monitoring will be used to measure 24h glucose profiles over 3-4 days prior to and following the acute exercise bout and again during the last week of the intervention. Continuous blood pressure monitoring will be used over 18-24 h, at the beginning and at the end of the 12 week-training.

Participants will take part in three postprandial metabolic studies: 1) before (A); 2) 18-24h after an acute exercise bout (B), and; 3) after 12-weeks of exercise training (C). Experiments will be conducted between 07:30 AM and 5:00 PM, following a 12 hr fast. Adipose tissue dietary fatty acid storage and partitioning of dietary fatty acids in skeletal muscles will be measured by the oral [18F-]-FTHA PET method. Changes in lean tissue mitochondrial function in vivo will be determined using magnetic resonance spectroscopy (MRS). Participants will complete Visit A (baseline), followed 7 to 14-days later by a pre-breakfast (9 AM) or pre-dinner (4PM) exhaustive glycogen lowering exercise bout. The following day (18-24h after the exercise bout), participants will return for a second metabolic visit (Visit B). Participants will then begin a 12-week supervised high-intensity interval training program, performed either only in the morning or only in the afternoon (9 AM vs. 4 PM), on every other day. At the end of the 12 weeks, and at least 48h after the last exercise bout, participants will return for their final metabolic visit (Visit C).

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetes:

  * Fasting plasma glucose: 6.1 to 6.9 mmol/L or
  * 2-hour plasma glucose post 75g OGTT: 7.8 to 11.0 mmol/L and
  * HbA1c: 6.0 to 6.4%
  * or Insulin resistant: glucose clearance rate ≤ 360 ml/kg/min as determined using the Oral Glucose Insulin Sensitivity Index at Time 120 min.
* BMI > 25 kg/m2
* To be willing and able to adhere to the specifications of the protocol;
* To have signed an informed consent document indicating that they understood the purpose of and procedures required for the study and were willing to participate in the study.

Exclusion Criteria:

* overt cardiovascular disease as assessed by medical history, physical exam, and abnormal ECG
* Treatment with any drug known to affect lipid or carbohydrate metabolism, except statins (to be stopped 3 weeks prior to study A), metformin or anti-hypertensive drugs (to be stopped 7 days prior to the studies);
* presence of liver or renal disease other than uncomplicated NASH or mild isolated proteinuria; uncontrolled thyroid disorder;
* Uncontrolled severe hypertension, systolic pressure ≥ 180 mm Hg or diastolic pressure ≥ 110 mm Hg;
* History of ischemic heart disease, tachyarrhythmia, QT interval prolongation, risk factors for torsade de pointes (eg hypokalemia), or taking any medication known to prolong the QT interval;
* History of serious gastrointestinal disorders (malabsorption, peptic ulcer, gastroesophageal reflux requiring surgery, etc.);
* Presence of a pacemaker;
* Having undergone a PET study or CT scan in the past year;
* Any contraindication to stopping statins for 3 months and stopping an anti-hypertensive medication and metformin for 7 days;
* smoking (>1 cigarette/day) and/or consumption of >2 alcoholic beverages per day;
* No blood donation two month prior the study;
* prior history or current fasting plasma cholesterol level > 7 mmol/l or fasting TG > 6 mmol/l.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Adipose tissue dietary fatty acid (DFA) partitioning | Measured 180 minutes, 240 minutes, 300 minutes and 360 minutes after liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using oral administration of [18F]-Fluoro-6-Thia-Heptadecanoic Acid (FTHA) during whole-body acquisition
Change in lean organ (heart, liver, skeletal muscle) DFA partitioning | Measured 180 minutes, 240 minutes, 300 minutes and 360 minutes after liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using oral administration of [18F]-Fluoro-6-Thia-Heptadecanoic Acid (FTHA) during whole-body acquisition
Change in skeletal muscle ATP fluxes in vivo | Measured 170 minutes before and 30 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using phosphorus-31 magnetic resonance spectroscopy.
Change in glucose control. | Measured continuously 2-3 days before and 2-3 days after first and final exercise session, after 12-week exercise intervention.
  Determined using continuous glucose monitoring and repeated blood samples obtained during metabolic visit.

SECONDARY OUTCOMES:
Change in adipose tissue nonesterified fatty acid (NEFA) metabolism. | Measured 150 minutes before and 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using [11C]-palmitate with dynamic PET acquisition
Change in lean organ (heart, liver, skeletal muscle) NEFA metabolism. | Measured 150 minutes before and 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using [11C]-palmitate with dynamic PET acquisition
Change in insulin sensitivity | Measured every 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined by measuring circulating glucose, NEFA, insulin and C-peptide following the liquid meal.
Change in dietary fatty acid oxidation | Measured every 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined by measuring breath [13C]-carbon dioxide enrichment.
Change in total substrate utilisation | Measured every 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using indirect calorimetry
Change in postprandial plasma NEFA turnover. | Blood sample collected every 60 min following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using continuous infusion of [7,7,8,8-2H]-palmitate.
Change in postprandial plasma glucose turnover | Blood sample collected every 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using continuous infusion of [1-3H]-glucose
Change in left ventricular function by Positron Emitting Positron (PET) ventriculography | Measured 150 minutes before and 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using [11C]-palmitate combined with ECG-gated cardiac dynamic PET acquisition.
Change in plasma distribution of DFA metabolites | Blood sample collected every 60 minutes following liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined using oral administration of [18F]-FTHA to quantify the incorporation of 18F-labeled fatty acids given with the liquid meal, into triglyceride-rich lipoproteins and NEFA.
Change in composition and activation status of immune cell subsets | Blood sample collected before and after liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined by extensive Fluorescence Activated cell Sorting (FACS) analysis
Change in plasma cytokine levels | Blood sample collected before and after liquid meal at baseline visit, 18-24hours after acute exercise bout and >48hours after final exercise bout (after 12 week intervention).
  Determined by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Denis P. Blondin, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
IPD from published manuscript will be provided upon reasonable request and dependent upon specific permission from the Comité d'éthique de la recherche du CIUSSS de l'Estrie-CHUS. In addition, the study protocol, statistical analysis plan and informed consent form may also be available upon reasonable request and approval from the Comité d'éthique de la recherche du CIUSSS de l'Estrie-CHUS.